CLINICAL TRIAL: NCT05201638
Title: A Multi-Center, Randomized, Double-Blinded Phase 3 Study to Evaluate the Efficacy, Safety, and Tolerability of IMU-838 Versus Placebo in Adults With Relapsing Multiple Sclerosis (ENSURE-2)
Brief Title: Study to Evaluate the Efficacy, Safety and Tolerability of IMU-838 in Patients With Relapsing Multiple Sclerosis
Acronym: ENSURE-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Immunic AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P3-IMU-838-RMS-02
Record Dates: First submitted 2021-12-13; First posted 2022-01-21 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IMU-838 (Experimental): IMU-838 (vidofludimus calcium), a small molecule inhibitor of DHODH.
  Formulation:
  Tablets with 15 or 30 mg IMU-838 for once daily oral intake in the morning.
  Interventions: Drug: IMU-838 tablets
- Placebo (Placebo Comparator): Matching placebo, as described for the test product, identical number of tablets as given for IMU-838.
  Interventions: Drug: Placebo matching IMU-838 tablets

INTERVENTIONS:
Drug: IMU-838 tablets — Patients are randomized to IMU-838 or placebo in ratio 1:1
  Other Names: Vidofludimus calcium
  Arms: IMU-838
Drug: Placebo matching IMU-838 tablets — Patients are randomized to IMU-838 or placebo in ratio 1:1
  Other Names: Placebo matching vidofludimus calcium
  Arms: Placebo

SUMMARY:
Multi-Center, Randomized, Double-Blinded Phase 3 Study to Evaluate the Efficacy, Safety, and Tolerability of IMU-838 versus Placebo in Adults with Relapsing Multiple Sclerosis (ENSURE-2)

DETAILED DESCRIPTION:
This study will be a multicenter, randomized, double-blind, placebo-controlled study with a blinded Main Treatment Period (MT) and an Open Label Period (OLE) to evaluate the efficacy, safety, and tolerability of IMU-838 in adult patients with RMS.

The study will consist of the following periods:

Screening Period: Approximately 28 days Main Treatment Period: 72 weeks (approximately 15 months) Open Label Extension Period: Up to approximately 8 years

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient (age ≥18 to ≤55 years).
* Patients with an established diagnosis of MS according to 2017 McDonald Criteria.
* Patients with RMS comprising of relapsing remitting MS (RRMS) and active secondary progressive MS, both defined according to Lublin criteria 1996 and 2014.
* Active disease as defined by Lublin 2014 evidenced prior to Screening by:

  1. At least 2 relapses in the last 24 months before randomization, or
  2. At least 1 relapse in the last 12 months before randomization, or
  3. A positive Gd+ MRI scan (brain and/or spine) in the last 12 months prior to randomization.
* Willingness and ability to comply with the protocol.
* Written informed consent given prior to any study-related procedure.

Exclusion Criteria:

* Patients with non-active secondary progressive MS and primary progressive MS.
* Any disease other than MS that may better explain the signs and symptoms, including history of complete transverse myelitis.
* Clinical signs or presence of laboratory findings suggestive for neuromyelitis optica (NMO) spectrum disorders or myelin oligodendrocyte glycoprotein (MOG)-IgG-associated encephalomyelitis
* Any active and uncontrolled coexisting autoimmune disease, other than MS (except for type 1 diabetes mellitus and inflammatory bowel disease)
* Use of experimental/investigational drug (with the exception of COVID-19 vaccines approved by emergency use authorization) and/or participation in drug clinical studies within 6 months prior to Screening
* Previous or current use of MS treatments lifelong, or within a pre-specified time period.
* Use of the pre-specified concomitant medications.
* Clinically significantly abnormal and pre-specified lab values.
* History of chronic systemic infections within 6 months before the date of informed consent.
* Diagnosis or suspected liver function impairment, which may cause fluctuating liver function tests during this study.
* Known history of nephrolithiasis or underlying condition with a strong association of nephrolithiasis.
* History or clinical diagnosis of gout.
* History or presence of any major medical or psychiatric illness
* Substantial medical condition that could create undue risk to the patient, could affect adherence with the study protocol or could undesirably affect study outcomes

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1050 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate efficacy of IMU-838 versus placebo based on time to first relapse | 72 weeks
  Survival analysis of time to first relapse, occurred after the start of study treatment administration and before the end of the double-blind period, censored at a maximum of 72 weeks.

SECONDARY OUTCOMES:
Effect of IMU-838 versus placebo on volume of new T2 lesions | 72 weeks
  To evaluate the effect of IMU-838 versus placebo on volume of new T2 lesions. Mean difference between IMU-838 and placebo in changes of the volume of new MRI T2 lesions over 24-weeks of treatment in the double-blind period.
Effect of IMU-838 versus placebo on disability progression | 72 weeks
  To evaluate the effect of IMU-838 versus placebo on disability progression. Survival analysis of time to 12-week confirmed disability progression, as measured on Expanded Disability Status Scale during the double-blind period, censored at maximum 72-weeks.
Effect of IMU-838 versus placebo on cognitive performance | 72 weeks
  To evaluate the effect of IMU-838 versus placebo on cognitive performance. Survival analysis of time to confirmed clinically relevant changes on Symbol Digit Modalities Test during the double-blind period, censored at maximum 72- weeks.
Effect of IMU-838 versus placebo on whole brain atrophy | 72 weeks
  To evaluate the effect of IMU-838 versus placebo on whole brain atrophy. Difference in the mean of the percentage change on the whole brain volume between IMU-838 and placebo during the 72-weeks double-blind period.
Safety of IMU-838 versus placebo | 72 weeks
  To evaluate safety and tolerability by assessment of occurrence of Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Fox, MD, Principal Investigator — Mellen Center for MS, Neurological Institute, Cleveland Clinic, Ohio
Locations (90):
- United States (7):
  - HonorHealth Research Institute - Bob Bove Neuroscience Institute, Scottsdale, Arizona
  - Neuro of Central Florida, Altamonte Springs, Florida
  - Healthcare Innovations, Coral Springs, Florida
  - Homestead Associates, Miami, Florida
  - Premier Clinical Research, Miami, Florida
  - Baptist Health Lexington, Nicholasville, Kentucky
  - Boston Clinical Trials, Boston, Massachusetts
- Armenia (2):
  - Heratsi Hospital Complex 1, Yerevan
  - Erebouni Medical Center, Yerevan
- Bosnia and Herzegovina (5):
  - UCC of Rep of Srpska, Banja Luka
  - Cantonal Hospital Bihac Dr. Irfan Ljubijankic, Bihać
  - University Clinical Center of Sarajevo, Sarajevo
  - University Clinical Center Sarajevo, Sarajevo
  - University Clinical Center Tuzla, Tuzla
- Astra Clinic, Tallinn, Estonia
- India (7):
  - Post-Graduation Institute of Medical Education and Research (PGIMER), Chandigarh
  - Fortis Memorial Research Institute, Gurugramam
  - Dr Ram Manohar Lohia Institute of Medical Sciences, Lucknow
  - All India Institute of Medical Sciences, New Delhi
  - GB Pant Institute of Postgraduate Medical Education and Research, New Delhi
  - SRI Guru Ram Das Institute of Medical Sciences and Research, Punjābi Bāgh
  - DKS PGI, Raipur
- Centro de Investig. Médicas, Lima, Peru
- Poland (10):
  - NZOZ Wielospecjalistyczna Poradnia Lekarska "Synapsis", Katowice
  - Neuro-Medic Janusz Zbrojkiewicz, Katowice
  - NZOZ Neuromed, Lublin
  - Indywidualna Praktyka Lekarska prof. Konrad Rejdak, Lublin
  - Instytut Zdrowia Boczarska, Oświęcim
  - NZOZ Hertmanowskiej, Plewiska
  - NZOZ Neuro-Kard, Poznan
  - Centrum Medyczne NeuroProtect, Warsaw
  - FutureMeds Warszawa Centrum, Warsaw
  - Centrum Med. Ibismed, Zabrze
- Romania (8):
  - SC Sana Monitoring SRL, Bucharest
  - Elias University Emergency Hospital, Bucharest
  - Clubul Sanatatii SRL, Campulung Muscel
  - Spitalul clinic CF Constanta, Constanța
  - Asociatia Comunitatea Oamenilor, Craiova
  - Aria Clinic SRL, Sibiu
  - Neuro Therapy, Timișoara
  - Spit Jud Branzeu TIM Neuro, Timișoara
- Serbia (10):
  - Klinicko bolnicki centar Dr Dragisa Misovic - Dedinje, Belgrade
  - Klinicko bolnicki centar Zvezdara, Belgrade
  - Opsta bolnica Medicinski sistem Beograd, Belgrade
  - Vojnomedicinska akademija, Belgrade
  - Univerzitetski Klinicki centar Kragujevac, Kragujevac
  - Univerzitetski Klinicki centar Nis, Niš
  - Hsptl Sveti Vracevi, Novi Kneževac
  - General Hospital Uzice, Užice
  - Klinicko Bolnicki centar Zemun, Zemun
  - Opsta bolnica Djordje Jovanovic Zrenjanin, Zrenjanin
- Turkey (Türkiye) (14):
  - Acibadem Adana Hospital, Adana
  - Adana Baskent Hospital, Adana
  - Baskent University Ankara Hospital, Ankara
  - Bezmialem Vakif University Hospital, Istanbul
  - T.C. Ministry of Health Istanbul Haseki Training and Research Hospital, Istanbul
  - Sancaktepe Sehit Prof.Dr. Ilhan Varank Training and Research Hospital, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Haydar Pasa Num. EAH, Istanbul
  - Kocaeli University Research and Application Hospital, Kocaeli
  - T.C. Ministry of Health Kutahya Provincial Directorate of Health Kutahya University of Health Sciences Evliya Celebi Training and Research Hospital, Kütahya
  - Manisa Celal Bayar University Hafsa Sultan Hospital, Manisa
  - 19 Mayis University Medical Faculty Hospital Health Application and Research Center, Samsun
  - Namik Kemal Uni Hospital, Tekirdağ
  - Zonguldak Bulent Ecevit University Health Practice and Research Hospital, Zonguldak
- Ukraine (23):
  - Communal noncommercial enterprise "First Cherkasy City Hospital", Cherkasy
  - MS Diagnosis Treatment Center, Cherkasy
  - Chernihiv City Hospital 4, Chernihiv
  - Municipal Institution "Dnipropetrovsk Regional Rehabilitation Hospital" of Dnipropetrovsk Regional Council", Dnipro
  - Ukrainian State Research Institute of Medico-Social Problems of Disability, Dnipro
  - "University Clinic" of Dnipro State Medical University, Department of Neurology, Dnipro
  - Dnipro City Hospital 6, Dnipro
  - Communal Non-Commercial Medical Enterprise "O.T.Bohayevskyi Kremenchuk City Hospital #1, Kremenchuk
  - State Institution "National Research Center for Radiation Medicine of the National Academy of Medical Sciences of Ukraine, Kyiv
  - 1 Private Clinic Medical Center, Kyiv
  - Dopomoga Plus medical center, Kyiv
  - Volyn Reg Clin Hospital, Lutsk
  - Lviv Regional Central Hospital, Lviv
  - 5 City Clin Hospital, Lviv
  - Communal institution "City Clinical Hospital №3" of Poltava City Council, Poltava
  - City Clinical Hospital 2, Rivne
  - Sumy Reg Clinical Hospital, Sumy
  - Salutem, Vinnytsia
  - LCC Medical center INET-09, Zaporizhzhya
  - Zaporizhia Med, Zaporizhzhya
  - Zaporizhia Regional Clinic Hospital, Zaporizhzhya
  - Zaporizhzhya City Hospital 6, Zaporizhzhya
  - Zaporizhzhya Hospital 9, Zaporizhzhya
- United Kingdom (2):
  - Royal Devon Uni NHS, Exeter
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No